CLINICAL TRIAL: NCT03986268
Title: The Effect of Vitamin D Replacement Therapy on Pathological Response in Breast Cancer Patients Treated With Neoadjuvant Therapy
Brief Title: Vitamin D Can Increase Pathological Response of the Breast Cancer Patients Treated With Neoadjuvant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Cetin Ordu, Assoc. Prof. Çetin Ordu, MD, Florence Nightingale Hospital, Istanbul
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2019-40016-06
Record Dates: First submitted 2019-05-26; First posted 2019-06-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Vitamin D Deficiency; Chemotherapy Effect; Pathology
Keywords: neoadjuvant treatment; Breast Cancer; Vitamin D3
MeSH Terms: conditions — Vitamin D Deficiency; Breast Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: The patients had measured a total of 25 OH vit D3 levels, previously treated with neoadjuvant therapy without replacement treatment with vitamine D3, as a control group, were planned to be compared with 30-50 patient in study groups at baseline and / or at the end of the treatment period. The pathological response rates of both groups were planned to be evaluated according to the molecular subtypes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): The patients measured a total of 25 OH vitamin D3 levels, initial, 3'th month and 6'th month of neoadjuvant therapy with replacement treatment with vitamin D3 at least weekly 50000 IU for eight weeks.
  Interventions: Drug: Vit D
- control group (Other): The patients had measured a total of 25 OH vitamin D3 levels, previously treated with neoadjuvant therapy without replacement treatment with vitamin D3.
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Vit D — The aim of this study is investigating pathologic response to neoadjuvant therapy if we give replacement therapy with vitamin D3 50.000 IU weekly dosage concurrent with chemotherapy in breast cancer patients.
  Other Names: Vitamin D3; cholecalciferol

SUMMARY:
The aim of the study is to evaluate the relationship between the vitamin D replacement and pathological response in patients undergoing neoadjuvant therapy according to different molecular sub types. Because of no study evaluating pathological response to neoadjuvant therapy with vitamin D replacement in patients with breast cancer.

DETAILED DESCRIPTION:
Calcitriol, a vitamin D metabolite, inhibits cell proliferation and pathways in invitro experiments. Vitamin D affects gene expression related to breast cancer and prevents cell differentiation, growth and angiogenesis . Low vitamin D may include a high risk of breast cancer, but there are also studies reporting that patients with low vitamin D levels at the time of diagnosis show more aggressive breast cancer course . Breast cells can produce vitamin D by taking part in the formation of 1,25 OH vit D3 in vitamin D synthesis as well as in kidney cells. Apoptosis can be caused by vitamin D receptors . There are very few studies on the effect of vitamin D replacement on breast cancer-related survival. There are studies reporting the incidence of fewer breast cancer with vitamin D replacement in contrast to there are studies showing the opposite .Patients achieved pathological complete response (PCR) with neoadjuvant therapy have been shown to have better survival. There are studies showing that they do not affect the PCR ratio related to the level of vitamin D in breast cancer patients receiving neoadjuvant chemotherapy. In one study, it was shown that it increases the response rate when given with bisphosphonate .There is no study evaluating pathological response to neoadjuvant therapy with vitamin D replacement in patients with breast cancer. The aim of the study is to evaluate the relationship between the vitamin D replacement and pathological response in patients undergoing neo-adjuvant therapy according to different molecular subtypes of biopsy-diagnosed breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer is confirmed by biopsy
* enough organ function,
* metabolically normal,
* eligible for neoadjuvant treatment
* The patients who were informed about the prerequisites with their consent

Exclusion Criteria:

* having metastatic disease
* having not operated from breast cancer after neoadjuvant treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
pathological complete response (PCR) | an average 24 weeks
  No residual tumor cells both in axilla and breast

SECONDARY OUTCOMES:
pathological complete response (PCR) relations with vitamin D levels | an average 24 weeks
  evaluating PCR in both axilla and breast in terms of levels of total 25 (OH) vitamin D at initial and after replacement vitamin D
pathological complete response (PCR) ratio regarding molecular sub types | an average 24 weeks
  evaluating PCR in both axilla and breast in terms of levels of total 25 (OH) vitamin D at initial and after replacement vitamin D according moleculary subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Çetin Ordu, Assoc. Prof, Principal Investigator — Gayrettepe FN Hospital; Fatma Aktepe, Prof, Study Director — Gayrettepe FN Hospital; Vahit Özmen, Prof, Study Chair — İstanbul FN hospital
Locations (1):
- İstanbul Florence Nightingale Hospital Breast Health Center, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The aim of the study was to evaluate the relationship between the vitamin D replacement and pathological response in patients undergoing biopsy-diagnosed neo-adjuvant therapy according to different molecular subtypes.

REFERENCES:
- [Result] Clark AS, Chen J, Kapoor S, Friedman C, Mies C, Esserman L, DeMichele A; I-SPY1 Investigators. Pretreatment vitamin D level and response to neoadjuvant chemotherapy in women with breast cancer on the I-SPY trial (CALGB 150007/150015/ACRIN6657). Cancer Med. 2014 Jun;3(3):693-701. doi: 10.1002/cam4.235. Epub 2014 Apr 9. PMID 24719175
- [Result] Shao T, Klein P, Grossbard ML. Vitamin D and breast cancer. Oncologist. 2012;17(1):36-45. doi: 10.1634/theoncologist.2011-0278. Epub 2012 Jan 10. PMID 22234628
- [Result] Rossi M, McLaughlin JK, Lagiou P, Bosetti C, Talamini R, Lipworth L, Giacosa A, Montella M, Franceschi S, Negri E, La Vecchia C. Vitamin D intake and breast cancer risk: a case-control study in Italy. Ann Oncol. 2009 Feb;20(2):374-8. doi: 10.1093/annonc/mdn550. Epub 2008 Aug 18. PMID 18711029
- [Result] Abbas S, Linseisen J, Chang-Claude J. Dietary vitamin D and calcium intake and premenopausal breast cancer risk in a German case-control study. Nutr Cancer. 2007;59(1):54-61. doi: 10.1080/01635580701390223. PMID 17927502
- [Result] Levi F, Pasche C, Lucchini F, La Vecchia C. Dietary intake of selected micronutrients and breast-cancer risk. Int J Cancer. 2001 Jan 15;91(2):260-3. doi: 10.1002/1097-0215(200002)9999:99993.3.co;2-r. PMID 11146455
- [Result] Viala M, Chiba A, Thezenas S, Delmond L, Lamy PJ, Mott SL, Schroeder MC, Thomas A, Jacot W. Impact of vitamin D on pathological complete response and survival following neoadjuvant chemotherapy for breast cancer: a retrospective study. BMC Cancer. 2018 Jul 30;18(1):770. doi: 10.1186/s12885-018-4686-x. PMID 30060745
- [Result] Zehnder D, Bland R, Williams MC, McNinch RW, Howie AJ, Stewart PM, Hewison M. Extrarenal expression of 25-hydroxyvitamin d(3)-1 alpha-hydroxylase. J Clin Endocrinol Metab. 2001 Feb;86(2):888-94. doi: 10.1210/jcem.86.2.7220. PMID 11158062
- [Derived] Ozkurt E, Ordu C, Ozmen T, Ilgun AS, Soybir G, Celebi F, Koc E, Ak N, Alco G, Kurt S, Agacayak F, Yavuz E, Tuzlali S, Ozmen V. Vitamin D Supplementation During Neoadjuvant Chemotherapy for Breast Cancer Improves Pathological Complete Response: A Prospective Randomized Clinical Trial. World J Surg. 2025 Jun;49(6):1396-1405. doi: 10.1002/wjs.12587. Epub 2025 Apr 14. PMID 40229998